CLINICAL TRIAL: NCT07022639
Title: Influence of Hospital Volume on Mortality and Length of Hospital Stay After Pancreatic Resection in Switzerland: A Retrospective National Registry Study
Brief Title: Influence of Hospital Volume on Mortality and Length of Hospital Stay After Pancreatic Resection in Switzerland
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Yanic Ammann, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: Hospital volume PR
Record Dates: First submitted 2025-05-26; First posted 2025-06-15 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Total pancreatectomy
  Interventions: Procedure: Total pancreatectomy
- Proximal pancreatectomy
  Interventions: Procedure: Proximal pancreatectomy
- Distal pancreatectomy
  Interventions: Procedure: Distal pancreatectomy

INTERVENTIONS:
Procedure: Total pancreatectomy — Total pancreatectomy for any kind of disease
  Groups: Total pancreatectomy
Procedure: Proximal pancreatectomy — Proximal pancreatectomy for any kind of disease
  Groups: Proximal pancreatectomy
Procedure: Distal pancreatectomy — Distal pancreatectomy for any kind of disease
  Groups: Distal pancreatectomy

SUMMARY:
The effect of centralisation measures on the operative outcomes after pancreatic resection in Switzerland has not been highlighted yet. This study aims to investigate the influence of the annual hospital specific case load of pancreatic resection on short-term postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with pancreatic resection in Switzerland between 2013 and 2022

Exclusion Criteria:

* incomplete case documentation
* age under 20 years
* other hospitals than general or surgical hospitals
* no index operation

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with pancreatic resection in Switzerland between 2013 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 6785 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Periprocedural
  The association between the hospital volume and the postoperative mortality Mortality Yes or No Hospital volume of pancreatic resection as marginal effect Association with GAM logistic regression

SECONDARY OUTCOMES:
Reoperation | Periprocedural
  The association between the hospital volume and the reoperation rate Reoperation Yes or No Hospital volume of pancreatic resection as marginal effect Association with GAM logistic regression
Length of hospital stay | Periprocedural
  The association between the hospital volume and the length of hospital stay Length of hospital stay in days Hospital volume of pancreatic resection as marginal effect Association with quantile regression
Sociodemographic trends | 2013 - 2022

CONTACTS AND LOCATIONS:
Locations (1):
- HOCH Health Ostschweiz, Kantonsspital St.Gallen, Sankt Gallen, St.Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No